CLINICAL TRIAL: NCT05976646
Title: Phase Ib/2a Drug-drug Interaction Study of a Combination of 45mg Dextromethorphan With 105 mg Bupropion (AUVELITY) as an Adjunctive Treatment for Buprenorphine/Naloxone for Opioid Use Disorder
Brief Title: Phase Ib/2a Drug-drug Interaction Study of a Combination of 45mg Dextromethorphan With 105 mg Bupropion
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HM20027635; 5UG1DA050207 (NIH)
Record Dates: First submitted 2023-07-24; First posted 2023-08-04 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Addiction; Opioid Use; Substance Use Disorders; Opioid Use Disorder
MeSH Terms: conditions — Behavior, Addictive; Substance-Related Disorders; Opioid-Related Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Subjects who are randomized to placebo will receive identical capsules to the test product at the same time periods noted above, administered orally.
  Interventions: Drug: Placebo
- Auvelity (Experimental): Orally-administered combination of dextromethorphan with Bupropion (trade name Auvelity)
  Interventions: Drug: Auvelity

INTERVENTIONS:
Drug: Placebo — Subjects who are randomized to placebo will receive identical capsules to the test product at the same time periods noted above, administered orally.
  Arms: Placebo
Drug: Auvelity — Orally-administered combination of 45 mg dextromethorphan with 105 mg Bupropion (trade name Auvelity). Auvelity will initially be administered orally once daily for three days. After 3 days on once daily AUVELITY, the participants will begin taking AUVELITY twice daily for 4 additional days as recommended in the FDA-approved prescribing information.
  Arms: Auvelity

SUMMARY:
The overall goal of this project is to collect initial human data on the effects of novel compounds on safety (interactions with an opioid drug, e.g., buprenorphine) and early efficacy signals (subjective effects on negative affect, craving, and opioid withdrawal) in OUD subjects currently in MOUD treatment with buprenorphine.

DETAILED DESCRIPTION:
The overall goal of this project is to collect initial human data on the effects of novel compounds on safety (interactions with an opioid drug, e.g., buprenorphine) and early efficacy signals (subjective effects on negative affect, craving, and opioid withdrawal) in OUD subjects currently in MOUD treatment with buprenorphine. The compound to be studied in this protocol will be a pre-configured combination of 45mg dextromethorphan with 105 mg Bupropion (AuvelityTM, hereafter referred as Auvelity). Notably, other NMDA receptor antagonists such as ketamine have also been shown to rapidly improve mood and reduce suicidality. OUD has also been linked to histories of trauma and syndromes of negative mood, where opioid use in many individuals was initially motivated by a desire to alleviate a negative mood state. Lastly, using the NIDA Phenotyping Battery, our group has also found negative emotionality to be part of a constellation of neurofunctional domains that are associated with SUD severity. Taken together, providing AUVELITY as an adjunctive treatment to buprenorphine could be an avenue to target crucial underlying mechanisms of OUD and improve OUD treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects between 18 - 65 years of age;
* Understand the study procedures and provide written informed consent in the English language.
* Meet current DSM-5 criteria for OUD, of at least moderate severity, currently engaged in MOUD treatment at a buprenorphine-naloxone sublingual film total daily dose ranging from 8mg/2mg to 24mg/6mg or buprenorphine sublingual tablet 5.7mg/1.4mg to 17.1/4.3 daily for at least 2 weeks at screening. Or on a stable dose of depot injectable buprenorphine for at least four months, with at least one week since last depot buprenorphine injection.
* Have a positive urine drug screen for buprenorphine during screening and upon presenting for the first laboratory day on the clinical research unit to document buprenorphine use;
* Quick Inventory of Depressive Symptomatology (16-Item) (QIDS-SR16) score of mild or greater (>6)
* Females must be non-pregnant and non-lactating. Additionally, for females with childbearing potential (ie., have not undergone sterilization via hysterectomy, bilateral tubal ligation, or bilateral oophorectomy, or at least 1 year post-menopausal), participants must agree to use an acceptable form of contraception during study participation and to continue its use for at least 30 days after the last dose of the study drug (e.g, abstinence, intrauterine device, hormonal implant, hormonal patch/ring/pill, condoms (male or female).

Exclusion Criteria:

* Contraindications for participation as determined by medical history and physical exam performed by study NP or study physician;
* Pregnant or nursing women;
* Baseline ECG with clinically significant abnormal conduction;
* Uncontrolled serious psychiatric or major medical disorder; including uncontrolled hypertension, seizure disorder, anorexia nervosa or bulimia, bipolar disorder, schizoaffective disorder, or schizophrenia;
* Taking antidepressant medications (tricyclic antidepressants, SSRIs, SNRIs, MAOIs), antibiotic linezolid, antiepileptics, or CNS stimulants (amphetamine, methylphenidate) within the two weeks prior to initiation of study medication
* History of adverse reaction or allergy to dextromethorphan or bupropion
* Current severe alcohol use disorder or current benzodiazepine use or recent (within last 3 months) discontinuation of alcohol with severe alcohol use disorder or discontinuation of benzodiazepines with severe benzodiazepine use disorder
* Current DSM-5 diagnosis of any psychoactive substance use disorder other than opioids, cocaine, marijuana, or nicotine, or mild or moderate alcohol use disorder. Diagnosis of mild to moderate use disorder for alcohol will not be considered exclusionary.
* Significant current suicidal or homicidal ideation (C-SSRS "yes" answers on questions 4 or 5) or a history of suicide attempt within the past 6 months.
* Any other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2023-09-18 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
Safety- as measured by heart rate | During each PK study visit from visit start to end, up to approximately 8 hours
  Heart rate (HR)
Safety- as measured by blood pressure | During each PK study visit from visit start to end, up to approximately 8 hours
  blood pressure
Safety- as measured by pulse oximetry | During each PK study visit from visit start to end, up to approximately 8 hours
  pulse oximetry
Safety- as measured by respiratory rate | During each PK study visit from visit start to end, up to approximately 8 hours
  respiratory rate
Safety- as measured by Adverse events | During each PK study visit from visit start to end, up to approximately 8 hours; and from baseline to end of study participation
  adverse events

SECONDARY OUTCOMES:
Buprenorphine PK | During each PK study visit from visit start to end, up to approximately 8 hours
  Plasma concentration-time profiles of buprenorphine and its metabolite norbuprenorphine

CONTACTS AND LOCATIONS:
Overall Officials: Frederick G Moeller, Principal Investigator — Virginia Commonwealth University
Locations (1):
- CARI Research Clinic- VCU Institute for Drug and Alcohol Studies, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-04-09): https://cdn.clinicaltrials.gov/large-docs/46/NCT05976646/ICF_000.pdf